CLINICAL TRIAL: NCT06636357
Title: Nitrous Oxide in the Treatment of Acute Suicidal Ideation
Acronym: NITOS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Sebastian Olbrich, Prof. Dr. med., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-01005
Record Dates: First submitted 2024-09-06; First posted 2024-10-10 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-10

CONDITIONS: Suicidality; EEG; Suicidal Ideation; Nitrous Oxide; Biomarkers / Blood; Biomarkers / Hair
Keywords: suicidality; nitrous oxide; suicidal ideation; depression
MeSH Terms: conditions — Suicidal Ideation; Depression | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50% nitrous oxide (N2O) plus 50% oxygen (Experimental): Patients will be treated with N20 (50% N2O combined with 50% oxygen) for 45 minutes. Both the study subject and the rater will be blinded to the treatment assignment.
  Interventions: Drug: 50% N2O plus 50% O2
- 50% oxygen plus 50% air (Placebo Comparator): Here, patients will be treated with 50% oxygen plus air for 45 minutes. Both the study subject and the rater will be blinded to the treatment assignment.
  Interventions: Drug: Oxygen (O2)

INTERVENTIONS:
Drug: 50% N2O plus 50% O2 — Inhalation of 50% N2O plus 50% O2 for 45 min
  Arms: 50% nitrous oxide (N2O) plus 50% oxygen
Drug: Oxygen (O2) — 50% O2 plus 50% air for 45 min
  Arms: 50% oxygen plus 50% air

SUMMARY:
The primary aim of the NITOS study is to investigate the potential rapid antisuicidal effects of N2O in the transdiagnostic treatment of suicidal ideation. On day 1, patients will receive either nitrous oxide (50% N2O balanced with oxygen) or placebo (50% oxygen balanced with air). Seven days after the first inhalation, a second inhalation will be performed. All patients will receive N2O at least once during this trial. While the first inhalation will be double-blind, only the patients but not the raters will be blinded to the second inhalation (day 8). For mechanism of action and prediction, a nested biomarker substudy will employ multimodal techniques including analysis of hair and blood samples, and EEG.

ELIGIBILITY:
Inclusion criteria:

* Ability to give written informed consent
* Moderate to severe suicidal ideation defined as a score ≥3 on the Montgomery-Asberg Depression Rating Scale (MADRS; Schmidtke et al., 1985) suicide item (item #10) as well as a self-report Beck Scale for Suicide Ideation (BSS; Kliem et al., 2017) items #4 plus #5 score ≥ 2
* Plasma homocysteine level ≤ 14 µmol/l

Exclusion criteria:

* Organic, including symptomatic, mental disorders (F00-F09; lifetime diagnosis)
* Schizophrenia, schizotypal and delusional disorders (F20-F29; lifetime diagnosis)
* Mental and behavioral disorders due to psychoactive substance use. Nicotine and cannabis will be ignored (F10-F19)
* Non-medical (i.e., recreational) use of inhalational N2O during the last 12 months
* Past intolerance or hypersensitivity to N2O
* Critical illness
* Severe cardiac disease
* Pregnancy or breastfeeding
* Pulmonary hypertension
* Chronic cobalamin or folate deficiency unless treated with folic acid and/or vitamin B12
* History or evidence of any other medical or neurological condition that would expose the subject to an undue risk of a significant adverse event as determined by the clinical judgment of the investigator
* Treatment with ketamine/esketamine during the last 4 weeks
* Treatment with opioid medications during the last 3 months
* Treatment with vagus nerve stimulation (VNS) or electroconvulsive therapy (ECT) within the last 3 months
* Recent (within the last 4 weeks) or current use of benzodiazepines in excess of 5 mg lorazepam or equivalent per day
* Finally, any other factors that, in the investigator's judgment, would unduly impact patient safety or compliance during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Beck Scale for Suicidal Ideation (BSS) | Day 0 to Day 2
  Change of BSS score between Day 0 and Day 2. Double-blind treatment with either N2O or placebo inhalation on Day 1.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS ) | Day 0 to Day 2
EEG changes associated with N2O / placebo inhalation | Day 1
  EEG will be performed before, during, and after inhalation
Suicide Visual Analog Scale (S-VAS) | Day 1
  Briefly, the S-VAS uses the phrase "urge to kill myself". Next to the phrase, the patient sees a line that is anchored on the left with the word "none" and on the right with the word "extreme" . Score ranges from 0 to 100.
Perceived Burdensomeness Visual Analog Scale (PB-VAS) | Day 1
  The PB-VAS uses the phrase "like a burden". Next to the phrase, the patient sees a line that is anchored on the left with the word "none" and on the right with the word "extreme" . Score ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kronenberg G, Bankwitz A, Provaznikova B, Muller M, Quednow BB, Seifritz E, Olbrich S. Inhalational nitrous oxide as a transdiagnostic approach for the treatment of suicidal ideation and suicidality in psychiatric inpatients: protocol for a double-blind randomised, controlled clinical single-centre trial. BMJ Open. 2025 Jul 16;15(7):e096825. doi: 10.1136/bmjopen-2024-096825. PMID 40669910